CLINICAL TRIAL: NCT07157098
Title: Asymmetrical High Flow Oxygen Versus Noninvasive Ventilation in Acute Hypercapnic Respiratory Failure
Acronym: HIFOLD2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 25-035
Record Dates: First submitted 2025-08-15; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Acute Hypercapnic Respiratory Failure
Keywords: acute hypercapnic respiratory failure; non-invasive ventilation; high-flow oxygen
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: Patients will go through three intervention steps, each with a different breathing support: asymmetrical high-flow nasal cannula (HFNC), non-invasive ventilation (NIV) using the standard NIV mask at the participating center, and NIV using a new mask design. Each step lasts 10 minutes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- All study patient (Experimental): Sequential respiratory support with 3 devices
  Interventions: Device: asymmetrical high-flow nasal cannula; Device: non-invasive ventilation with standard mask; Device: non-invasive ventilation with a new mask

INTERVENTIONS:
Device: asymmetrical high-flow nasal cannula — high-flow nasal oxygen therapy via asymmetrical nasal prongs
Device: non-invasive ventilation with standard mask — non-invasive ventilation with standard oronasal mask, clinically used in the participting site
Device: non-invasive ventilation with a new mask — non-invasive ventilation with a new mask design, with under-nose, bridge-free design

SUMMARY:
NIV is a life-saving treatment for people with breathing failure and carbon dioxide (CO2) retention. It helps remove this waste gas from the lungs and reduces the effort needed to breathe. However, the standard masks used for NIV can become uncomfortable over time, which may lead patients to stop using them. Stopping treatment can be dangerous and may cause breathing problems to worsen. That's why finding devices that are more comfortable and possibly more effective is very important. This study aims to take a first step in that direction.

This is the first study comparing new devices designed to help people with chronic CO2 buildup during breathing flare-ups. Devices tested include a new type of asymmetrical nasal cannula for high-flow oxygen therapy and a new mask called OptiNIV, which has a comfortable design that may help remove more CO2.

These devices will be compared to standard NIV masks currently used in hospitals. Outcome of interests include their effects on the effort needed to breathe, on how much CO2 is cleared, and on how comfortable they are.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with acute hypercapnic respiratory failure
* Admitted to the intensive care unit
* Being treated with either high-flow oxygen treatment or non-invasive ventilation

Exclusion Criteria:

* Clinical instability - defined as the presence of one of the followings: respiratory rate > 40 breaths/minute, SpO2 < 80%, active broncho-pleural fistula, Glasgow Coma Scale < 8, mean arterial pressure below 60 mmHg despite usage of vasopressors
* Requiring immediate need of endotracheal intubation, according to the judgement of the attending physician
* Contraindications of monitoring with electrical impedance tomography (e.g. pacemaker, chest wall burns wounds limiting electrode placement).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Power of Breathing | Minute 10, 20, and 30
  A marker of the patient's work of breathing. Calculated by thickening fraction of the diaphragm, multiplied by the respiratory rate.

SECONDARY OUTCOMES:
Ventilatory Ratio | Minute 10, 20, and 30
  A marker of ventilation efficiency. Calculated from carbon dioxide level (in this case, obtained from transcutaneous capnography) and minute ventilation (in this case, obtained from electrical impedance tomography)
Patient's comfort | Minute 10, 20, and 30
  Obtained from a visual analog scale from 1 to 10, with 10 indicating the highest comfort
Patient's subjective shortness of breath | Minute 10, 20, and 30
  Obtained from a visual analog scale from 1 to 10, with 10 indicating the worst shortness of breath

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The datasets generated and/or analyzed during the current study are not publicly available due participant confidentiality, according to the REB, but are available from the corresponding author on reasonable request.